CLINICAL TRIAL: NCT00123513
Title: Images of a Healthy Worksite-Preventing Weight Gain in the Workplace
Brief Title: Workplace-Sponsored Program to Reduce Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Diana Fernandez, Associate Professor, Department of Community and Preventive Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 196; R01HL079511 (NIH)
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Obesity; Cardiovascular Diseases
MeSH Terms: conditions — Obesity; Cardiovascular Diseases | interventions — Diet; Exercise; Environment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Worksite intervention for obesity prevention
  Interventions: Behavioral: Diet; Behavioral: Exercise; Behavioral: Environment
- 2 (No Intervention): Control group

INTERVENTIONS:
Behavioral: Diet — Environmental changes in the food and physical activity environment. Cafeteria and vending machine changes, food brought from home, walking routes, and awareness building.
  Other Names: Obesogenic environment
  Arms: 1
Behavioral: Exercise — Increase routing physical activity, walking routes, stairs intervention, etc.
  Arms: 1
Behavioral: Environment — Cafeteria and vending machine changes and identification of opportunities of physical activity.
  Arms: 1

SUMMARY:
The purpose of this study is to design a comprehensive nutrition and physical activity strategy to gain a broad understanding of the social and cultural role of food and physical activity among workers. Perspectives on innovative interventions that are socially feasible and culturally acceptable will also be obtained. Health lifestyle promotion interventions addressing portion control, healthy nutrition, and increasing physical activity will be tested.

DETAILED DESCRIPTION:
BACKGROUND:

Broad, population-based approaches are needed to stop or reverse the rise in obesity prevalence. According to the World Health Organization, obesity prevention can be achieved by promoting a healthy diet and a physically active lifestyle. A partnership with the Eastman Kodak Company has been developed to test a worksite intervention for obesity prevention in Rochester, New York.

DESIGN NARRATIVE:

The overall goal of this study is to design a comprehensive nutrition and physical activity strategy based on participatory research to promote a healthy lifestyle and to stop the shift of the population body mass index (BMI) curve to the right. Six pairs of worksites will be randomized to either an intervention or control group. Two cross-sectional samples of employees within each worksite will be measured at baseline and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Full-time employees in good health

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3938 (Actual)
Dates: Start 2004-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
BMI | Measured at baseline and Year 2

SECONDARY OUTCOMES:
Number of serving of fruits and vegetables | Measured at baseline and Year 2
Number of steps a day | Measured at baseline and Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Isabel D. Fernandez, MD, MPH, PhD, Principal Investigator — University of Rochester
Locations (1):
- Eastman Kodak Company, Rochester, New York, United States